CLINICAL TRIAL: NCT02657733
Title: Comparison Study Between Nellcor Respiration Rate Technology (RRoxi) and Masimo Acoustic Respiration Rate (RRa)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oridion (Industry)
Collaborators: Herzog Hospital (Other)
Responsible Party: Sponsor
Organization: Medtronic - MITG (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 10144939
Record Dates: First submitted 2015-11-09; First posted 2016-01-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Respiratory Conditions for Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteers (Other): Respiration rate will be measured using several medical devices: Radical-7, Capnostream20p and Nellcor Bedside Respiratory Patient Monitoring System
  Interventions: Device: Radical-7; Device: Nellcor™ Bedside Respiratory Patient Monitoring System; Device: Capnostream 20p

INTERVENTIONS:
Device: Radical-7 — Comparison between 3 different monitors that measure respiratory rate. The participant is connected to 3 monitors at the same time.
  Radical-7- measures respiratory rate according to acoustic respiratory rate (RRa).
Device: Nellcor™ Bedside Respiratory Patient Monitoring System — Comparison between 3 different monitors that measure repiratory rate. The participant is connected to 3 monitors at the same time.
  Nellcor™ Bedside Respiratory Patient Monitoring System - measures respiratory rate according to oximetry respiration rate (RRoxi).
Device: Capnostream 20p — Comparison between 3 different monitors that measure respiratory rate. The participant is connected to 3 monitors at the same time. Capnostream 20p- measures respiratory rate according to Capnography (RRetco2).

SUMMARY:
Respiration rate is a critical vital sign that provides early detection of respiratory compromise and patient distress. Continuous monitoring of respiration rate is performed in patients under different clinical conditions, including post-surgery or different respiratory diseases. Clinician observation, pulse oximetry, and capnography are used individually or in combination to monitor ventilation during sedation and on post-surgical patients. The American Society of Anesthesiologists mandates the monitoring of respiration by measuring end tidal carbon dioxide (RRetco2) during procedural sedation and anesthesia. Other techniques for respiration rate measurement include different technologies such as acoustic respiratory rate (RRa). The aim of this study is to compare the accuracy of RRetco2 and RRa under certain respiratory conditions.

ELIGIBILITY:
Inclusion Criteria:

* Without Clinical diagnosis of chronic obstructive pulmonary disease (COPD)
* Without Clinical diagnosis of heart disease.

Exclusion Criteria:

* Want to be excluded
* Breathing difficulties
* Unabling or unwilling to follow the protocol.
* Contact allergy to the adhesive neck sensor.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The influence of different breathing rates (normal breathing, tachypnea, and bradypnea) on the accuracy of respiratory rate in breaths per minute as measured by the tested devices compared to a reference device. | 6 hours
  Respiratory rate will be measured with the monitors (Radical-7 device, Nellcor device, Capnostream20p device) and recorded in the following units: Breath/minute. Differences in accuracy as compared to the reference device and differences in percentage of time in which the device was accurate will be analyzed offline.

SECONDARY OUTCOMES:
The influence of hearing or performing noises on the accuracy of respiratory rates (in breaths per minute) as measured by the tested devices compared to a reference device. | 6 months
  Respiratory rate will be measured with the monitors (Radical-7 device ,Nellcor device, Capnostream20p device) in breaths per minute. Differences in accuracy as compared to the reference device and differences in percentage of time in which the device indicated respiratory rate values will be analyzed offline.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Eisenberg, MD, Principal Investigator — Herzog Hospital
Locations (1):
- Herzog Hospital, Jerusalem, Israel